CLINICAL TRIAL: NCT02227095
Title: Exercise & Overweight Children's Cognition
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Georgia (Other); San Francisco State University (Other)
Responsible Party: Principal Investigator, Catherine Davis, Professor of Pediatrics, Physiology & Graduate Studies, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: R01HL087923 (NIH); R01HL087923 (NIH)
Record Dates: First submitted 2014-04-23; First posted 2014-08-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- After-school exercise program (Experimental): 40 min/day vigorous aerobic games after school
  Interventions: Behavioral: Exercise; Behavioral: After-school program
- Sedentary after-school program (Active Comparator): Attention-control condition similar to experimental condition with the exception of exercise
  Interventions: Behavioral: After-school program

INTERVENTIONS:
Behavioral: Exercise — Heart rate monitors worn by each child at each session
  Other Names: Aerobic training
  Arms: After-school exercise program
Behavioral: After-school program — Supervised recreational program with token economy

SUMMARY:
This research focuses on overweight, sedentary children whose health, cognition, and academic performance are therefore at risk, and who may be particularly responsive to exercise interventions.

This study will determine whether regular exercise per se (i.e. compared to attention control, or placebo, condition) benefits children's cognition and achievement, and will provide insight into neural mechanisms. A substudy will examine exercise-induced changes in brain structure.

Provision of comprehensive evidence for the benefits of exercise on children's health may reduce barriers to vigorous physical activity programs during a childhood obesity epidemic by persuading policymakers, schools and communities that time spent in physical activity enhances, rather than detracts from, learning.

DETAILED DESCRIPTION:
An ancillary study adding cardiometabolic outcome measures was added (R01HL087923-02S1, http://projectreporter.nih.gov/project_info_description.cfm?aid=7880457&icde=20104167)

ELIGIBILITY:
Inclusion Criteria:

* 8-11 years of age
* Overweight or obese (BMI-for-age >= 85th percentile)
* Able to participate in exercise testing and intervention

Exclusion Criteria:

* Medical condition or medications that would interfere with measurements
* Participation in weight control or formal exercise program outside physical education that meets more than 1 day/week
* T-score > 75 on the BRIEF Behavior Regulation scale to avoid program disruption

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2008-05; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Planning Scale scores | Baseline, 8 months, one-year follow-up
  The Cognitive Assessment System provides an individually administered standardized psychological assessment of executive function
Change in functional MRI | Baseline, 8 months
  Change in blood-oxygenation level dependent (BOLD) signal reflecting brain activation during executive function tasks

SECONDARY OUTCOMES:
Change in BMI | Baseline, 8 months, one-year follow-up
  BMI and BMI z-score, per current norms, will be calculated
Change in adiposity | Baseline, 8 months, one-year follow-up
  Percent fat via whole-body dual-energy x-ray absorptiometry
Change in aerobic fitness | Baseline, 8 months, one-year follow-up
  VO2 peak via treadmill test
Change in Tower of London scores | Baseline, 8 months, one-year follow-up
  Individually administered standardized psychological assessment of executive function
Change in teacher ratings of classroom behavior | Baseline, 8 months
  Behavior Rating Inventory for Executive Functions-Teacher form
Change in academic achievement | Baseline, 8 months, one-year follow-up
  Woodcock-Johnson Test of Achievement III
Change in performance on executive function tasks | Baseline, 8 months
  Antisaccade and flanker tasks - error rates, interference effect

OTHER OUTCOMES:
Change in physical activity outside the program | Baseline, 8 months, one-year follow-up
  Youth Risk Behavior Survey questions at all 3 timepoints, accelerometry at baseline and 8 months
Attendance to the interventions | 8 months
Average heart rate during the exercise intervention | 8 months
  Polar heart rate monitors will be worn by each child in the exercise intervention and downloaded after each session. Average heart rate during the session will be recorded daily. The mean for each child over the intervention period will be computed.
Points earned during the intervention | 8 months
  Points earned for expected behavior will be recorded daily for each child that attends the intervention. Points are redeemed for small prizes weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Davis, PhD, Principal Investigator — Medical College of Georgia, Georgia Regents University; Jennifer E McDowell, PhD, Principal Investigator — University of Georgia
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States

REFERENCES:
- [Result] Krafft CE, Schwarz NF, Chi L, Weinberger AL, Schaeffer DJ, Pierce JE, Rodrigue AL, Yanasak NE, Miller PH, Tomporowski PD, Davis CL, McDowell JE. An 8-month randomized controlled exercise trial alters brain activation during cognitive tasks in overweight children. Obesity (Silver Spring). 2014 Jan;22(1):232-42. doi: 10.1002/oby.20518. Epub 2013 Sep 10. PMID 23788510
- [Result] Krafft CE, Pierce JE, Schwarz NF, Chi L, Weinberger AL, Schaeffer DJ, Rodrigue AL, Camchong J, Allison JD, Yanasak NE, Liu T, Davis CL, McDowell JE. An eight month randomized controlled exercise intervention alters resting state synchrony in overweight children. Neuroscience. 2014 Jan 3;256:445-55. doi: 10.1016/j.neuroscience.2013.09.052. Epub 2013 Oct 3. PMID 24096138
- [Result] Krafft CE, Schaeffer DJ, Schwarz NF, Chi L, Weinberger AL, Pierce JE, Rodrigue AL, Allison JD, Yanasak NE, Liu T, Davis CL, McDowell JE. Improved frontoparietal white matter integrity in overweight children is associated with attendance at an after-school exercise program. Dev Neurosci. 2014;36(1):1-9. doi: 10.1159/000356219. Epub 2014 Jan 21. PMID 24457421
- [Result] Schaeffer DJ, Krafft CE, Schwarz NF, Chi L, Rodrigue AL, Pierce JE, Allison JD, Yanasak NE, Liu T, Davis CL, McDowell JE. An 8-month exercise intervention alters frontotemporal white matter integrity in overweight children. Psychophysiology. 2014 Aug;51(8):728-33. doi: 10.1111/psyp.12227. Epub 2014 May 5. PMID 24797659
- [Result] Schaeffer DJ, Krafft CE, Schwarz NF, Chi L, Rodrigue AL, Pierce JE, Allison JD, Yanasak NE, Liu T, Davis CL, McDowell JE. The relationship between uncinate fasciculus white matter integrity and verbal memory proficiency in children. Neuroreport. 2014 Aug 20;25(12):921-5. doi: 10.1097/WNR.0000000000000204. PMID 24949818
- [Derived] Williams CF, Bustamante EE, Waller JL, Davis CL. Exercise effects on quality of life, mood, and self-worth in overweight children: the SMART randomized controlled trial. Transl Behav Med. 2019 May 16;9(3):451-459. doi: 10.1093/tbm/ibz015. PMID 31094443